CLINICAL TRIAL: NCT07237828
Title: Drainage Removal After Reverse-Sequence Endoscopic Nipple-Sparing Mastectomy With Direct-to-Implant Prepectoral Breast Reconstruction on Postoperative Safety and Patient Satisfaction : A National Multicenter, Open, Randomized Controlled Study
Brief Title: Drain Removal on Postoperative Safety and Patient Satisfaction in R-E-NSM With Prepectoral DIBR
Acronym: DRAIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Du Zhenggui (Other)
Collaborators: The First Affiliated Hospital of Shanxi Medical University (Other); West China Fourth Hospital, Sichuan University (Unknown); Bethune Hospital of Shanxi Medical University (Unknown); The First Hospital of Jilin University (Other); Shanxi Province Cancer Hospital (Other); Suining Central Hospital (Other); The Second Affiliated Hospital of Kunming Medical University (Other); Zhengzhou Central Hospital (Other); Deyang People's Hospital (Other); Suzhou Municipal Hospital (Other); Chengdu Fifth People's Hospital (Other); Hunan University of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Zhengzhou University (Other); The Fourth People's Hospital of Sichuan Province (Unknown); China-Japan Union Hospital, Jilin University (Other); Guangzhou First People's Hospital (Other); Xinjiang Medical University Affiliated Cancer Hospital (Unknown); Fujian Medical University Union Hospital (Other); Central Hospital of Taiyuan (Unknown); West China Tianfu Hospital of Sichuan University (Unknown)
Responsible Party: Sponsor-Investigator, Du Zhenggui, Clinical Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025(440)
Record Dates: First submitted 2025-09-20; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Minimal invasive surgery; Nipple-sparing mastectomy; Endoscopic surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Remove drainage tubes on postoperative day 5
  Interventions: Procedure: Drain Removal Timing After Endoscopic Breast Reconstruction Surgery
- Control group (No Intervention): Remove drainage tubes when the daily drainage volume is less than 30 ml/day for two consecutive days after surgery.

INTERVENTIONS:
Procedure: Drain Removal Timing After Endoscopic Breast Reconstruction Surgery — The optimal timing for earlier or later removal of drainage tubes after endoscopic breast reconstruction surgery.
  Arms: Intervention group

SUMMARY:
Breast cancer is a malignant tumor that seriously threatens the health of women, with an increasing incidence rate. The current main treatment methods include multidisciplinary diagnosis and treatment such as surgery, radiotherapy, chemotherapy, and endocrine therapy, among which surgery is the key. Postoperative care is also very important. Traditional breast surgery requires long-term placement of drainage tubes after the operation. However, long-term placement of drainage tubes increases the incidence of postoperative complications such as infection and delayed wound healing, prolongs hospital stays, increases economic burden, and also affects the aesthetic outcome. Our team has innovatively adopted the "reverse-sequence" endoscopic nipple-sparing-mastectomy with direct-to-implant breast reconstruction. This method is highly efficient and safe, with no incisions on the surface of the breast, reducing the risk of incision dehiscence and the probability of flap ischemia and necrosis. Based on this, our team proposes to appropriately relax the drainage criteria and remove the drainage tube earlier under the premise of ensuring the sterility of the effusion, and preliminary findings show that patients have better postoperative aesthetic outcomes, with a lower incidence of flap infection, ischemia, and necrosis than expected, and the degree of breast deformation caused by radiotherapy is also reduced. However, there is still controversy over the pros and cons of drainage criteria. Some scholars believe that strict drainage criteria can reduce the risk of infection and implant displacement, and plastic surgeons are more concerned about the impact of long-term tube placement on aesthetic outcomes and quality of life. Currently there is a lack of large sample, multicenter, randomized controlled studies to provide high - level evidence. Therefore, our team plans to conduct a national multicenter, open, randomized controlled study to compare the advantages and disadvantages of the two drainage methods under the premise of not reducing postoperative surgical and oncological safety, in order to explore the optimal timing for drain removal and improve patients' satisfaction with the reconstructed breast.

DETAILED DESCRIPTION:
This study is a multicenter, open, randomized controlled trial. Prior to group allocation, participants were stratified by axillary lymph node dissection. The proportion of patients undergoing axillary lymph node dissection is 25%, while the proportion of patients not undergoing axillary lymph node dissection is 75%. Following stratification, participants within each stratum were randomized in a 3:1 ratio to the intervention or control groups. The target sample size is 379 participants, comprising 95 in the ALND group (71 intervention, 24 control) and 284 in the non-ALND group (213 intervention, 71 control).

An interim analysis will occur 1 year after study initiation and 1 month post-enrollment completion. Final analysis follows 5-year postoperative follow-up for all participants. Categorical variables will be analyzed using chi-square or Fisher's exact tests; continuous variables via t-tests, ANOVA, or non-parametric alternatives (Mann-Whitney/Kruskal-Wallis) as appropriate. Survival outcomes will employ Kaplan-Meier curves with log-rank testing.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-70 years (inclusive);
* Patients scheduled for unilateral or bilateral reverse-sequence endoscopic nipple-sparing- mastectomy with immediate prepectoral direct-to-implant breast reconstruction, with the option of concurrent contralateral endoscopic breast augmentation;
* Patients with preoperative pathological confirmation of carcinoma in situ, invasive cancer, or those undergoing prophylactic mastectomy;
* Patients with a maximum tumor diameter≤5 cm (before/after neoadjuvant chemotherapy), and no clinical or radiological evidence of nipple, skin, chest wall invasion, or distant metastasis;
* BMI < 40 kg/m²;
* Implant volume < 600 mL;
* Patients who are able and willing to sign the informed consent form.

Exclusion Criteria:

* History of breast surgery within 1 year prior to this operation (excluding VABB and biopsy);
* Tumor invasion of the skin, pectoralis major muscle, chest wall, or nipple-areola complex;
* Advanced tumor stage (M1);
* Breast cancer during pregnancy or lactation;
* Scars below the nipple level and a history of previous radiotherapy;
* Patients with severe comorbidities before surgery, poorly controlled diabetes, immunodeficiency, or poor general condition that cannot tolerate surgery;
* HbA1c > 7.5%;
* Active smoking history (≥20 cigarettes per day);
* Intraoperative flap burns, intraoperative nipple excision; postoperative complications such as infection, flap ischemia, or surgical cavity bleeding within 1-4 days after surgery; or other causes leading to incisions on the surface of the breast; patients who undergo nipple excision within 1 month after surgery should be excluded from the study;
* Currently participating in other clinical studies that may affect participation in this trial.
* Refusal to sign the informed consent form.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2032-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Aesthetic outcome evaluation--BREAST-Q scores | Preoperative (baseline), 3-month postoperative
  The Satisfaction with Breasts module of BREAST-Q questionnaire is utilized to assess patient-reported aesthetic outcomes. Transformed scores range from 0 to 100, with higher scores indicating better outcomes. Both raw questionnaire scores and standardized transformed scores will be documented, along with pre- to postoperative differences in transformed scores

SECONDARY OUTCOMES:
Drainage tube indwelling duration | Perioperative
  The duration of drainage tube indwelling refers to the total time from the postoperative insertion of the drainage tube to its removal, measured in days
Quality of Life--EORTC Quality of Life scores | 14 days postoperative and 3 months postoperative
  EORTC Scores are a series of questionnaires developed by the European Organisation for Research and Treatment of Cancer (EORTC) to assess the health-related quality of life (HRQoL) of cancer patients. These questionnaires are widely used in clinical trials and clinical practice to help evaluate treatment outcomes and patients' quality of life. The scoring range is from 0 to 100. A higher score in the functional domains indicates better functioning, while a higher score in the symptom domains indicates more severe symptoms.
wound care | 3 months postoperative
  The differences in the number of dressing changes and wound care procedures.
Complications | 3 months, 1 year and 2 years postoperative
  Skin flap thermal injury, skin flap ischemia/necrosis, nipple and areola complex(NAC) ischemia/necrosis, surgical site infection, incision dehiscence, surgical site bleeding or hematoma, seroma needing repeated aspiration or drain reinsertion, capsular contracture, prosthesis outline appearance, rippling, implant displacement, implant loss, readmission
Aesthetic outcome evaluation--BREAST-Q scores | 2 years postoperative
  The Satisfaction with Breasts module of BREAST-Q questionnaire is utilized to assess patient-reported aesthetic outcomes. Transformed scores range from 0 to 100, with higher scores indicating better outcomes. Both raw questionnaire scores and standardized transformed scores will be documented, along with pre- to postoperative differences in transformed scores
Quality of Life--BREAST-Q scores | Preoperative (baseline), 3 months and 2 years postoperative
  The Psychosocial Well-Being, Sexual Well-Being, and Physical Well-Being of the Chest modules of BREAST-Q questionnaire are used to evaluate quality of life (QoL) outcomes. Transformed scores range from 0 to 100, with higher values indicating better outcomes. Both raw questionnaire scores and standardized transformed scores will be recorded, along with pre- to postoperative differences in transformed scores
Surgical margin involvement | 2-3 weeks postoperative after paraffin-embedded pathological report available
  Surgical margin involvement was defined as ink on tumor on postoperative paraffin-embedded pathological examination
The total volume of drainage | Perioperative
  The volume of drainage refers to the total amount of fluid drained from the time of tube placement to the time of tube removal, measured in milliliters.
Aesthetic outcome evaluation--Harris score | 2-year postoperative
  The Harris score was used to record the subjective judgment of symmetry of the reconstructed breast compared to the contralateral breast. The results were categorized as excellent (treated breast nearly identical to untreated breast), good (treated breast slightly different than untreated), fair (treated breast clearly different than untreated), and poor (treated breast seriously distorted).
Aesthetic outcome evaluation--Ueda score | 2-year postoperative
  Doctor-reported aesthetic outcomes will be evaluated by three professional breast surgeons using the Ueda scale, based on postoperative photographs. Scores range from 0 to 10 points, with higher values indicating better results. The categorized as follows: Excellent (≥9 points), Good (7-8 points), Fair (5-6 points), Poor (≤4 points). Both raw scores and categorizations will be documented
Local Recurrence-Free Survival(LRFS) | 2-year postoperative and 5-year postoperative
  The time interval from initiation of treatment to the first recurrence at the primary tumor site.If local recurrence appears, record the time and location of recurrence
Disease-Free Survival(DFS) | 2-year postoperative and 5-year postoperative
  The period from treatment initiation to any disease recurrence (local, regional, or distant) or death.If above event appears, record the time and disease location.
Overall Survival(OS) | 2-year postoperative and 5-year postoperative
  The time from treatment initiation (or diagnosis) to death from any cause. If death appears, record the time and reason.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, SiChuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data via the request portal. All IPD requests should be emailed to Dr. Zhenggui Du, the general project leader, and will be evaluated by Dr. Du and the head of the collaborating organization to decide whether to approve.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of relevant research outputs, such as academic papers and books.
Access Criteria: When a request has been approved, the investigator will provide access to the de-identified individual patient-level data in the data management platform (Electronic Data Capture, EDC). A signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing the requested information. Additionally, all users will need to accept the terms and conditions of the data management platform to gain access.
URL: https://dct.meddb.cn/login_index

REFERENCES:
- [Background] Feng Y, Xie Y, Liang F, Zhou J, Yang H, Qiu M, Zhang Q, Liu Y, Liang P, Du Z. Twenty-four-hour discharge of patients after endoscopic nipple-sparing mastectomy and direct-to-implant breast reconstruction: safety and aesthetic outcomes from a prospective cohort study. Br J Surg. 2024 Jan 3;111(1):znad356. doi: 10.1093/bjs/znad356. No abstract available. PMID 37991082
- [Background] Zhou J, Xie Y, Liang F, Feng Y, Yang H, Qiu M, Zhang Q, Chung K, Dai H, Liu Y, Liang P, Du Z. A novel technique of reverse-sequence endoscopic nipple-sparing mastectomy with direct-to-implant breast reconstruction: medium-term oncological safety outcomes and feasibility of 24-h discharge for breast cancer patients. Int J Surg. 2024 Apr 1;110(4):2243-2252. doi: 10.1097/JS9.0000000000001134. PMID 38348883
- [Background] Yang H, Liang F, Xie Y, Qiu M, Du Z. Single axillary incision reverse-order endoscopic nipple/skin-sparing mastectomy followed by subpectoral implant-based breast reconstruction: Technique, clinical outcomes, and aesthetic results from 88 preliminary procedures. Surgery. 2023 Sep;174(3):464-472. doi: 10.1016/j.surg.2023.05.037. Epub 2023 Jul 7. PMID 37422354
- [Background] Zhang S, Xie Y, Liang F, Wang Y, Wen N, Zhou J, Feng Y, Liu X, Lv Q, Du Z. Video-assisted Transaxillary Nipple-sparing Mastectomy and Immediate Implant-based Breast Reconstruction: A Novel and Promising Method. Aesthetic Plast Surg. 2022 Feb;46(1):91-98. doi: 10.1007/s00266-021-02527-6. Epub 2021 Aug 23. PMID 34424367
- [Background] Jia-Jian C, Nai-Si H, Jing-Yan X, Ben-Long Y, Guang-Yu L, Gen-Hong D, Zhi-Min S, Jiong W. Current Status of Breast Reconstruction in Southern China: A 15 Year, Single Institutional Experience of 20,551 Breast Cancer Patients. Medicine (Baltimore). 2015 Aug;94(34):e1399. doi: 10.1097/MD.0000000000001399. PMID 26313786
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338